CLINICAL TRIAL: NCT06595706
Title: A Phase 1, Randomised, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety and Pharmacokinetics of Lucid-21-302 in Healthy Adult Participants
Brief Title: Evaluating the Safety and Pharmacokinetics of Multiple Ascending Doses of Lucid-21-302 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huge Biopharma Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Quantum Biopharma (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Lucid-21-302-002
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Heathy Participants

STUDY DESIGN:
Intervention Model Description: 2 MAD cohorts. Each MAD cohort will enroll 8 participants randomized 6 active:2 placebo to receive multiple doses of Lucid-21-302.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lucid-21-302 (Experimental): Multiple ascending dose cohorts
  Interventions: Drug: Lucid-21-302
- Placebo (Placebo Comparator): Multiple ascending dose cohorts
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lucid-21-302 — Capsule containing a small molecule inhibitor of hypercitrullination
  Arms: Lucid-21-302
Drug: Placebo — Capsule containing only Silicified Microcrystalline Cellulose
  Arms: Placebo

SUMMARY:
This study aims to determine the safety and pharmacokinetics of multiple ascending doses of Lucid-21-302 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 and ≤60 years (inclusive), with BMI >18.0 and <32.0 kg/m2 and body weight ≥50.0 kg. Social smokers consuming less than 10 cigarettes per week, with a negative cotinine test at screening and Day -1 will be allowed.
2. Participant is judged by the Investigator to be in generally good health on the basis of medical history, physical examination, or clinical laboratory results during the screening.
3. Pulse between 45 and 100 beats per minute (bpm) in supine position at screening (inclusive)
4. Supine systolic BP between 90 and 160 mmHg, diastolic BP between 50 and 95 mmHg inclusive, at screening. For the purpose of qualifying any given participant for study participation, out-of-range vital signs may be repeated once.
5. Ability to consume standard meals and the ability to fast for at least ten hours.
6. Agree not to have a tattoo or body piercing until the end of the study.
7. Agree not to receive the COVID-19 vaccination or other vaccination from seven days prior to the study drug dose until seven days after study drug administration in the study.
8. Must not be pregnant, breastfeeding (non-lactating), or planning pregnancy.
9. Female participants must have negative serum hCG pregnancy test at screening and negative urine test a check-in.
10. Females of childbearing potential who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomised at least 6 months prior to the first study drug administration) must be willing to use one of the following acceptable contraceptive methods throughout the study and for at least 1 month after the last study drug administration:

    a. Simultaneous use of intrauterine contraceptive device with or without hormone release system placed at least 4 weeks prior to the first study drug administration; and a condom for the male partner. Oral contraceptives are not allowed.
11. Females of non-childbearing potential must be:

    1. Post-menopausal (absence of menses for at least 12 months prior to the first study drug administration) with confirmation of the post menopausal status by documented FSH level ≥40 mIU/mL; or
    2. Surgically sterile (complete hysterectomy or bilateral oophorectomy at least 3 months prior to the first study drug administration).
12. Female participants must be willing not to donate ova for 90 days after the last dose
13. Male participants who are not vasectomised for at least 6 months prior to dosing and who are sexually active with a female partner of childbearing potential must be willing to use one of the following acceptable contraceptive methods from the first dose and for 90 days after the last dose:

    a. Simultaneous use of condom and hormonal contraceptive (e.g., oral, patch, depot injection, implant, vaginal ring, intrauterine device) or non-hormonal intrauterine device used for at least 4 weeks prior to sexual intercourse for the female partner;
14. All male participants (including men who have had a vasectomy) must agree to use a condom from the first dose and for 90 days after the last dose.
15. Male participants must be willing not to donate sperm for 90 days after the last dose.
16. Willing and able to adhere to all study requirements, including willingness to remain in the study unit for the entire duration of the confinement period.
17. Participant has a good venous access.
18. Able to understand the study procedures and provide signed and dated participant informed consent form (ICF) to participate in the study prior to screening.

Exclusion criteria:

1. History of any clinically significant gastrointestinal, renal, hepatic (except cholecystectomy), neurologic, hematologic, endocrine, oncologic, pulmonary (except resolved childhood astma), immunologic, or cardiovascular disease or other condition which would jeopardize safety or impact validity of results (in the opinion the Investigator); history of common medical conditions such as depression (non-hospitalised, but potentially medicated in the past), migraine or Gilbert syndrome will not be allowed unless the exemption will be provided by the Investigator.
2. Participant has any documented clinically significant infection, injury, or illness within 1 month prior to screening.
3. Participant has any documented history of, or currently active, seizure disorder (any seizure including infantile seizures), or history of clinically significant head injury based on the opinion of the Investigator.
4. Participants who have a history of surgery within 6 months prior to screening, or who have a plan of surgery during the study. Small surgeries such as dental operation, biopsies and non-invasive surgeries may be allowed at Investigator discretion.
5. Liver function test results elevated more than 1.5-fold above the upper limit of normal (ULN) for gamma glutamyl transferase (GGT), bilirubin (total, conjugated and unconjugated), alkaline phosphatase (ALP), aspartate aminotransferase (AST) or alanine aminotransferase (ALT). Volunteers with ALP and/or ALT/AST above the limits specified may be included, at the discretion of the Investigator, if the levels are unaccompanied by clinical signs and are determined to be normal variants; Testing for any out-of-range values may be repeated once at the discretion of the Investigator.
6. A calculated creatinine clearance of < 60 mL/minute at Screening according to the equation using Cockcroft and Gault.

   Testing for any out-of-range laboratory tests values may be repeated once at the discretion of the Investigator.
7. Participant has an active malignancy of any type or has been diagnosed with cancer within 5 years prior to screening (excluding squamous or basal cell carcinoma of the skin).
8. Any laboratory test results deemed clinically significant by the Investigator or positive test serology test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen and antibody at screening.

   Testing for any out-of-range laboratory tests values may be repeated once at the discretion of the Investigator.
9. History of inherent cardiac abnormalities based on the opinion of the Investigator.
10. Clinically significant ECG abnormalities in supine position defined at the Investigator discretion (Fridericia's corrected QT interval [QTcF] >440 ms for males and >460 ms for females), PR >210 ms, QRS interval > 120 ms at screening.

    Testing for any out-of-range values may be repeated once at the discretion of the Investigator.
11. Clinically significant bradycardia or tachycardia in supine position defined at the Investigator discretion as resting heart rate (HR) <44 bmp or > 101 bpm, respectively.

    Testing for any out-of-range values may be repeated once at the discretion of the Investigator.
12. Positive urine drug screen, urine cotinine and alcohol breath test and at screening or check-in.

    Testing may be repeated once at the discretion of the Investigator.
13. History or presence of food allergies and dietary restrictions, which, in the opinion of the Investigator, would prevent the participant from participating in the study.
14. Known history or presence of severe allergic reactions (e.g., anaphylactic reactions, angioedema), which, in the opinion of the Investigator, would prevent the participant from participating in the study.
15. Participants with a score ≥ 10 for the Modified Patient Health Questionnaire (PHQ-9) or the Modified Generalized Anxiety Disorder 7-item (GAD-7) or Columbia Suicide Severity Rating Scale (C-SSRS)
16. History of significant drug abuse (as per Investigator's discretion) such as cocaine, phencyclidine (PCP), crack, opioid derivatives including heroin, and amphetamine derivatives within 1 year prior to screening and throughout the study.
17. Use of marijuana (directly or indirectly) within 90 days prior to drug administration and during the course of the study.
18. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit that exceeds 14 units of alcohol per week (1 unit = 150 mL of wine, 375 mL of mid strength beer, or 30 mL of distilled alcohol 40%).
19. Use of medications for the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or participant safety (e.g., topical drug products without significant systemic absorption):

    1. Prescription medications (except for allowed contraceptives) within 14 days prior to the first dose until end of the study;
    2. Monoamine oxidase inhibitors (MAOIs) within 28 days prior to dosing;
    3. Over-the-counter products and natural health products (including herbal remedies such as St. John's wort, homeopathic and traditional medicines), and antacid preparations within 30 days prior to the first dose up to end of study. Vitamins and dietary supplements used as nutritional supplements in non-therapeutic doses (judged by the qualified Investigator or designee) must be stopped at least 14 days before dosing and during the study.
    4. Any drugs known to induce or inhibit hepatic and renal drug metabolism within 30 days prior to the first dose and during the study.
    5. Use of any enzyme-modifying drugs and/or other products, including strong inhibitors of cytochrome P450 (CYP) enzymes (e.g., cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (e.g., barbiturates, carbamazepine, glucocorticoids, phenytoin, St. John´s Wort, and rifampicin) in the previous 30 days before study drug administration.
20. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days (or a minimum of 5 half-lives, whichever is longer) prior to the first dose, administration of a biological product in the context of a clinical research study within 90 days prior to the first dose, or concomitant participation in an investigational study involving no drug or device administration.
21. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 56 days prior to Day -1.
22. Any reason which, in the opinion of the Investigator, would prevent the participant from participating in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-09-28 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and relationship of Adverse Events (AEs) | Up to 15 days
  Safety Outcome Measure
Incidence of Serious AEs (SAEs) and suspected unexpected SAEs | Up to 15 days
  Safety Outcome Measure
Number of discontinuations due to AEs | Up to 15 days
  Safety Outcome Measure
Clinically significant changes from baseline in complete blood count | Up to 15 days
  Safety blood test measured by a laboratory using a reference range
Clinically significant changes from baseline in blood coagulation | Up to 15 days
  Safety blood test measured by a laboratory using a reference range
Clinically significant changes from baseline in blood biochemistry | Up to 15 days
  Safety blood test measured by a laboratory using a reference range
Clinically significant changes from baseline in urinalysis | Up to 15 days
  Safety urine test measured by a laboratory using a reference range
Clinically significant changes from baseline in physical exam | Up to 15 days
  Safety Outcome Measure, clinical exam performed by a licensed physician
Clinically significant changes from baseline in systolic blood pressure | Up to 15 days
  Safety Outcome Measure, measured in mmHg
Clinically significant changes from baseline in diastolic blood pressure | Up to 15 days
  Safety Outcome Measure, measured in mmHg
Clinically significant changes from baseline in heart rate | Up to 15 days
  Safety Outcome Measure, measured in beats per minute
Clinically significant changes from baseline in respiratory rate | Up to 15 days
  Safety Outcome Measure, measured in breaths per minute
Clinically significant changes from baseline in tympanic temperature | Up to 15 days
  Safety Outcome Measure, measured in degrees Celcius
Clinically significant changes from baseline in 12-lead electrocardiogram (ECG) | Up to 15 days
  Safety Outcome Measure, measured using a standard ECG machine
Clinically significant changes from baseline in patient health questionnaire (PHQ-9) | Up to 15 days
  Safety Outcome Measure, PHQ-9 is a depression scale with scores ranging from 0 to 27 with higher scores indicating more depressive symptoms
Clinically significant changes from baseline in generalized anxiety disorder questionnaire (GAD7) | Up to 15 days
  Safety Outcome Measure, GAD7 is an anxiety scale with scores ranging from 0 to 21 with higher scores indicating more anxiety symptoms
Clinically significant changes from baseline in Columbia suicide severity rating scale (C-SSRS) | Up to 15 days
  Safety Outcome Measure, C-SSRS is an assessment tool that measures suicidal ideation and behavior. It consists of ten yes or no questions with yes answers indicating more thoughts of suicidality.
Clinically significant changes from baseline in neurological exam | Up to 15 days
  Safety Outcome Measure, neurological exam performed by a licensed physician

SECONDARY OUTCOMES:
AUC from time zero to 24 hours | Day1 (pre-dose to 24 hours post-dose)
  PK characteristic on Day 1
AUC from time zero to the last non-zero concentration | Day1 (pre-dose to 24 hours post-dose)
  PK characteristic on Day 1
Maximum concentration (Cmax) | Day1 (pre-dose to 24 hours post-dose)
  PK characteristic on Day 1
Time to maximum concentration (Tmax) | Day1 (pre-dose to 24 hours post-dose)
  PK characteristic on Day 1
AUC from time zero to the end of the dosing period | Day 4 (pre-dose to 24 hours post-dose)
  PK characteristic on Day 4
AUC from time zero to the last non-zero concentration | Day 4 (pre-dose to 24 hours post-dose)
  PK characteristic on Day 4
Minimum concentration (Cmin) | Day 4 (pre-dose to 24 hours post-dose)
  PK characteristic on Day 4
Maximum concentration (Cmax) | Day 4 (pre-dose to 24 hours post-dose)
  PK characteristic on Day 4
Time to maximum concentration (Tmax) | Day 4 (pre-dose to 24 hours post-dose)
  PK characteristic on Day 4
AUC from time zero to the last non-zero concentration | Day 7 (pre-dose to 48 hours post-dose)
  PK characteristic on Day 7
Maximum concentration (Cmax) | Day 7 (pre-dose to 48 hours post-dose)
  PK characteristic on Day 7
Time to maximum concentration (Tmax) | Day 7 (pre-dose to 48 hours post-dose)
  PK characteristic on Day 7
Minimum concentration (Cmin) | Day 7 (pre-dose to 48 hours post-dose)
  PK characteristic on Day 7
AUC from time zero to infinity | Day 7 (pre-dose to 48 hours post-dose)
  PK characteristic on Day 7
Average concentration at steady state (Css ave) | Day 7 (pre-dose to 48 hours post-dose)
  PK characteristic on Day 7
AUC from time zero to the end of the dosing period | Day 7 (pre-dose to 48 hours post-dose)
  PK characteristic on Day 7
Residual area | Day 7 (pre-dose to 48 hours post-dose)
  PK characteristic on Day 7
Elimination half-life | Day 7 (pre-dose to 48 hours post-dose)
  PK characteristic on Day 7
Elimination rate constant | Day 7 (pre-dose to 48 hours post-dose)
  PK characteristic on Day 7
Apparent clearance of drug at steady state | Day 7 (pre-dose to 48 hours post-dose)
  PK characteristic on Day 7
Apparent volume of distribution at steady state | Day 7 (pre-dose to 48 hours post-dose)
  PK characteristic on Day 7
AUC accumulation ratio | Day 1 to Day 7
  PK characteristic
Maximum concentration (Cmax) accumulation ratio | Day 1 to Day 7
  PK characteristic
Trough concentration | Day 2 to Day 7
  PK characteristic

CONTACTS AND LOCATIONS:
Locations (1):
- Cmax Clinical Research, Adelaide, Maryland, Australia

IPD SHARING:
Plan to Share IPD: No